CLINICAL TRIAL: NCT04487145
Title: DPART Study: Dihydroartemisinin-Piperaquine in the Context of Antiretroviral Therapy
Brief Title: Dihydroartemisinin-Piperaquine in the Context of Antiretroviral Therapy
Acronym: DPART
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: Yale University (Other); Makerere University (Other); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 18-26978; 2R01HD068174-06A1 (NIH)
Record Dates: First submitted 2020-07-17; First posted 2020-07-27 (Actual); Results first posted 2025-03-14 (Actual); Last update posted 2025-03-14 (Actual); Status verified 2025-02

CONDITIONS: Drug-Drug Interaction; HIV Infection
Keywords: Drug drug interaction; HIV; malaria; dihydroartemisinin; piperaquine; lopinavir; ritonavir; efavirenz; dolutegravir; Children
MeSH Terms: conditions — HIV Infections; Malaria

STUDY DESIGN:
Intervention Model Description: This is an open-label prospective pharmacokinetic and safety study of DP and 3 different ART regimens (EFV-, LPV/r- and DTG-based ART) in non-malaria-infected 1) HIV-infected children and 2) HIV uninfected children not on ART (controls).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (7):
- HIV-infected children on EFV-based ART (E3) (Experimental): 30 HIV-infected children age 3 - 10 years on EFV-based ART for at least 10 days will take standard 3 consecutive once-daily oral doses of DP (20/120mg tablets) based on weight per 2015 WHO guidelines for DP. The brand name Duocotexin will be used.
  Interventions: Drug: Dihydroartemisinin-piperaquine
- HIV-infected children on DTG-based ART (D3) (Experimental): 30 HIV-infected children age 11 - 17 years on DTG-based ART for at least 10 days will take standard 3 consecutive once-daily oral doses of DP (20/120mg tablets) based on weight per 2015 WHO guidelines for DP. The brand name Duocotexin will be used.
  Interventions: Drug: Dihydroartemisinin-piperaquine
- HIV-infected children on LPV/r-based ART (L3) (Experimental): 30 HIV-infected children age 3 - 10 years on LPV/r-based ART for at least 10 days will take standard 3 consecutive once-daily oral doses of DP (20/120mg tablets) based on weight per 2015 WHO guidelines for DP. The brand name Duocotexin will be used.
  Interventions: Drug: Dihydroartemisinin-piperaquine
- HIV-uninfected children (C3a) (Active Comparator): 30 HIV-uninfected children age 3-10 years not on ART will take standard 3 consecutive once-daily oral doses of DP (20/120mg tablets) based on weight per 2015 WHO guidelines for DP. The brand name Duocotexin will be used. PK samples are collected after the 3rd dose. Control group for E3 and L3.
  Interventions: Drug: Dihydroartemisinin-piperaquine
- HIV-uninfected children (C3b) (Active Comparator): 30 HIV-uninfected children age 11-17 years not on ART will take standard 3 consecutive once-daily oral doses of DP (20/120mg tablets) based on weight per 2015 WHO guidelines for DP. The brand name Duocotexin will be used. Control group for D3.
  Interventions: Drug: Dihydroartemisinin-piperaquine
- HIV-uninfected children (C1) (Active Comparator): 20 HIV-uninfected children age 3-10 years not on ART will take standard 3 consecutive once-daily oral doses of DP (20/120mg tablets) based on weight per 2015 WHO guidelines for DP. The brand name Duocotexin will be used. PK samples are collected after the 1st dose. Control group for L1.
  Interventions: Drug: Dihydroartemisinin-piperaquine
- HIV-infected children on LPV/r-based ART (L1) (Experimental): 20 HIV-infected children age 3 - 10 years on LPV/r-based ART for at least 10 days will take one oral dose DP (20/120mg tablets) based on weight per 2015 WHO guidelines for DP. The brand name Duocotexin will be used
  Interventions: Drug: Dihydroartemisinin-piperaquine

INTERVENTIONS:
Drug: Dihydroartemisinin-piperaquine — It is expected that efavirenz (EFV), lopinavir/ritonavir (LPV/r), and/or dolutegravir (DTG) will alter DP exposure.
  Other Names: DP; Duocotexin; Eurartesim; DHA-PQ

SUMMARY:
Open-label prospective intensive pharmacokinetic study of dihydroartemisinin-piperaquine (DP) in HIV-infected children on efavirenz (EFV)-, lopinavir/ritonavir (LPV/r)-, or dolutegravir (DTG)-based antiretroviral therapy (ART) and HIV-uninfected children not on ART. All children will be malaria-uninfected at the time of enrollment.

DETAILED DESCRIPTION:
The primary goal of the study is to assess the pharmacokinetics (PK) and safety of DP in the setting of co-administration with first-line ART regimens (EFV-, LPV/r- or DTG-based ART) in children without malaria. Up to 190 children will be enrolled in one of the 5 groups: 1, HIV-infected children age 3 - 10 years on LPV/r-based ART (n=20 for signal dose DP, 30 standard 3-dose DP). 2, HIV-infected children age 3 - 10 years on EFV-based ART (n=30), 3, HIV-infected children age 11 - 17 years on DTG-based ART (n=30), 4, HIV-uninfected children age 3-10 years (standard 3-dose DP, n=20 for PK sampling after the 1st dose DP, n=30 for sampling after the 3rd dose DP), 5, HIV-uninfected children age 11-17 years (n=30 children receiving 3-dose DP).

HIV-infected participants will be enrolled from the Baylor Uganda Center of Excellence on the Mulago Hospital Complex, Kampala, Uganda. HIV-uninfected participants will be enrolled from Masafu General Hospital (MGH) complex in Busia, and other clinics in the surrounding area. DP weight-based dosing will follow World Health Organization (WHO) Treatment Guidelines for uncomplicated malaria (April 2015). All HIV-infected participants must be stabilized (i.e. no change in regimen for at least 10 days) on EFV, LPV/r, or DTG + 2 nucleoside reverse transcriptase inhibitors (NRTI). HIV-infected children on LPV/r will be enrolled in two Phases: Phase I participants (Group L1) will receive a single dose of DP to determine the magnitude (PK and safety) of the interaction before 3 doses are evaluated, Phase II participants (Group L3) will receive a 3-dose DP regimen (which consists of 3 days of a once daily DP dose). Phase I results will inform Phase II dosing, as a lower dose of DP over 3 days may be warranted. Phase II will not begin until PK and safety results from Phase I are evaluated. Participants in L1 and L3 will be encouraged to participate sequentially in Phase I and Phase II separated by a minimum 42-day washout period; however different children may be enrolled for the 2 phases. Weight-based dose of dihydroartemisinin-piperaquine (DP): 5- <8kg, 20+160mg; 8- <11kg, 30+240mg; 11- <17kg, 40+320mg; 17- <25kg, 60+480mg; 25- <36kg, 80+640mg; 36- <60kg, 120+960mg; 60-<80kg, 160+1280mg; >80kg, 200+1600mg.

Subjects will undergo an intensive PK study sampling design, which entails multiple venous blood collections in a smaller sample of individuals to accurately estimate drug exposure over time. These studies will be conducted in both HIV-infected and HIV-uninfected participants and will allow the researchers to investigate dihydroartemisinin (DHA) and piperaquine (PQ) PK exposure in the context of EFV-, LPV/r- and DTG-based ART in HIV-uninfected children. Comparisons will be based on an intensive PK design for DP area under the concentration-time curve (AUC) estimations. A sample size of 20 children/adolescents will be needed in groups L1 and C1. A sample size of 30 will be needed for each of the other arms (D3, E3, L3, C3a, and C3b). Sampling will occur up to day 42 in the 3-dose groups given the long half-life of PQ and for 14 or 28 days in the single dose groups. The generation of an AUC will permit robust comparisons so that results will inform treatment guidelines and policy.

ELIGIBILITY:
Inclusion Criteria:

All participants:

* Agreement to come to clinic for all follow-up PK and safety evaluations
* Provision of informed consent.

HIV-infected participants:

* Residency within 30km of Mulago Hospital.
* Confirmed HIV infection (confirmed positive rapid HIV test or HIV RNA as per
* Ugandan guidelines).
* On stable EFV-, LPV/r- or DTG-based ART for at least 10 days prior to enrollment.
* Age 3 - 10 years if on EFV-based ART or LPV/r-based ART.
* Age 11 - 17 years if on DTG-based ART.

HIV-uninfected participants:

* Residency within 30km of Masafu General Hospital
* Confirmed HIV negative test (confirmed positive rapid HIV test or HIV RNA as
* per Ugandan guidelines)
* Age 3 - 17 years.

Exclusion Criteria:

* History of significant comorbidities such as malignancy, active tuberculosis or
* other active WHO stage 4 disease
* Receipt of any medications known to affect CYP450 metabolism (except ART)
* within 14 days of study enrolment (see 4.2.1)
* Hemoglobin < 7.0 g/dL
* Current malaria infection or recent treatment with antimalarials within 28 days of
* enrolment.
* Asymptomatic parasitemia detected by microscopy or rapid diagnostic test (RDT)
* History of side effects with DP
* Prior history of cardiac disease (personal or family), baseline corrected QT intervals (QTc) >450msec, or
* receipt of any cardiotoxic drugs or those known to prolong QT intervals History of
* significant comorbidities such as malignancy, active tuberculosis or other WHO
* stage 4 disease
* Weight < 6kg
* HIV-infected females on DTG-based ART and age 13-17 years who are pregnant
* or of childbearing potential and do not agree to consistent and reliable
* contraception.

The following medications are disallowed within 3 weeks prior to receiving study drug:

* Carbamazepine
* Clarithromycin
* Erythromycin (oral)
* Ketoconazole
* Phenobarbital
* Phenytoin
* Rifabutin
* Rifampicin
* Halofantrine
* Any other medication known to significantly affect CYP450 metabolism.
* Grapefruit juice should be avoided during the study due to its potential effects on CYP3A4.

Ages: 3 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 194 (Actual)
Dates: Start 2020-11-23 (Actual); Primary Completion 2022-04-11 (Actual); Study Completion 2022-04-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Francesca Aweeka, Principal Investigator — University of California, San Francisco; Sunil Parikh, Principal Investigator — Yale University; Norah Mwebaza, Principal Investigator — Makerere University; Adeodata Kekitiinwa, Study Chair — Baylor College of Medicine Children's foundation Uganda
Locations (2):
- Uganda (2):
  - Masafu General Hospital (MGH) at Busia District, Eastern Uganda, Masafu, Busia
  - Baylor-Uganda Center of Excellence on Mulago Hospital Complex and Masafu General Hospital, Kampala

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Single dose study only enrolled 20 children in L1 and 20 in C1 to evaluate the safety in the context of DP and LPV/r drug-drug interaction, only one dose of DP was given in the treatment group (L1). None of those children were included in the 5 groups in the 3-dose full study. So this is not a two-period design.
Period: Single-dose Study for Safety Evaluation
Arm/Group | HIV-uninfected Children (C3a) | HIV-infected Children on LPV/R-based ART (L3) | HIV-infected Children on EFV-based ART (E3) | HIV-uninfected Children (C3b) | HIV-infected Children on DTG-based ART (D3) | HIV-uninfected Children (C1) | HIV-infected Children on LPV/R-based ART (L1)
Started | 0 | 0 | 0 | 0 | 0 | 20 | 20
Completed | 0 | 0 | 0 | 0 | 0 | 20 | 20
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: 3-dose Study
Arm/Group | HIV-uninfected Children (C3a) | HIV-infected Children on LPV/R-based ART (L3) | HIV-infected Children on EFV-based ART (E3) | HIV-uninfected Children (C3b) | HIV-infected Children on DTG-based ART (D3) | HIV-uninfected Children (C1) | HIV-infected Children on LPV/R-based ART (L1)
Started | 30 | 30 | 31 | 32 | 31 | 0 | 0
Completed | 30 | 30 | 30 | 30 | 30 | 0 | 0
Not Completed | 0 | 0 | 1 | 2 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | HIV-infected Children on EFV-based ART (E3) | HIV-infected Children on DTG-based ART (D3) | HIV-infected Children on LPV/R-based ART (L3) | HIV-uninfected Children (C3a) | HIV-uninfected Children (C3b) | HIV-uninfected Children (C1) | HIV-infected Children on LPV/R-based ART (L1) | Total
Number analyzed (Participants) | 30 | 30 | 30 | 30 | 30 | 20 | 20 | 190
Age, Continuous [Median (Inter-Quartile Range); unit: years] — DTG age upper limit is 17 years, which could be up to 17.9 years as long as the age did not reach 18 years.
  years | 7.9 [6.6 to 9.1] | 15.3 [13.5 to 17.2] | 7.1 [6.1 to 8.7] | 7.4 [6.0 to 8.7] | 14.7 [13.5 to 16.3] | 6.2 [4.3 to 8.4] | 6.5 [5.0 to 9.0] | 8.7 [6.4 to 13.2]
Sex: Female, Male [Count of Participants; unit: Participants]
  sex: Female | 19 | 13 | 15 | 11 | 13 | 13 | 8 | 92
  sex: Male | 11 | 17 | 15 | 19 | 17 | 7 | 12 | 98
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 30 | 30 | 30 | 30 | 30 | 20 | 20 | 190
  White | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Uganda | 30 | 30 | 30 | 30 | 30 | 20 | 20 | 190
Weight [Median (Inter-Quartile Range); unit: kg] | 21.4 [18.0 to 25.9] | 48.7 [38.8 to 53.4] | 19.0 [17.4 to 22.4] | 23.6 [21.5 to 27.8] | 42.7 [36.8 to 53.2] | 20.1 [16.2 to 24.1] | 18.9 [16.9 to 27.6] | 25.0 [18.9 to 37.7]

OUTCOME MEASURES:

1. Primary Outcome: AUC0-42day in 3-dose Study
Description: AUC 0-day42 (from time 0 to 42 days) for piperaquine
Time Frame: 42 days
Population: Only five arms in 3-dose study. because C1 and L1 were only for single-dose study to evaluate safety, and those participants were not in 3-dose study,
Measure: Geometric Mean (95% Confidence Interval); unit: hr.ug/mL
Arm/Group | HIV-infected Children on EFV-based ART (E3) | HIV-infected Children on DTG-based ART (D3) | HIV-infected Children on LPV/R-based ART (L3) | HIV-uninfected Children (C3a) | HIV-uninfected Children (C3b)
Number analyzed (Participants) | 30 | 30 | 30 | 30 | 30
hr.ug/mL | 4.47 [3.83 to 5.22] | 14.9 [12.0 to 18.2] | 49.7 [41.7 to 59.2] | 14.6 [12.7 to 16.7] | 19.2 [16.6 to 22.2]

2. Primary Outcome: QTcF in 3-dose Study
Description: Safety of 3-dose DP regimens determined via-assessment of mean change in QT intervals from baseline; Here we reported mild adverse event defined as QTc F change>30ms but <60ms from baseline.
Time Frame: 42 days
Population: We only have five arms in 3-dose study. because C1 and L1 were only for single-dose study to evaluate safety. those participants were not in 3-dose study,
Measure: Count of Participants; unit: Participants
Arm/Group | HIV-infected Children on EFV-based ART (E3) | HIV-infected Children on DTG-based ART (D3) | HIV-infected Children on LPV/R-based ART (L3) | HIV-uninfected Children (C3a) | HIV-uninfected Children (C3b)
Number analyzed (Participants) | 30 | 30 | 30 | 30 | 30
Participants | 0 | 3 | 8 | 2 | 2

3. Primary Outcome: AUC0-day28 in 3-dose Study
Description: Area under concentration -time curve from pre-3rd dose to day 28
Time Frame: day 2-28
Population: We only have five arms in phase 2. because C1 and L1 were only for phase 1 safety evaluation. those participants were not in phase 2 study,
Measure: Geometric Mean (90% Confidence Interval); unit: hr.ug/mL
Arm/Group | HIV-infected Children on EFV-based ART (E3) | HIV-infected Children on DTG-based ART (D3) | HIV-infected Children on LPV/R-based ART (L3) | HIV-uninfected Children (C3a) | HIV-uninfected Children (C3b)
Number analyzed (Participants) | 30 | 30 | 30 | 30 | 30
hr.ug/mL | 4.33 [3.71 to 5.06] | 12.7 [10.3 to 15.7] | 41.6 [34.8 to 49.9] | 12.5 [10.9 to 14.4] | 16.4 [14.1 to 19.1]

4. Primary Outcome: Cmax for Piperaquine in 3-dose Study
Description: maximal piperaquine concentration post the 3rd dose (day 2-42)
Time Frame: day 2-28
Population: as for outcome 2
Measure: Geometric Mean (90% Confidence Interval); unit: ng/mL
Arm/Group | HIV-infected Children on EFV-based ART (E3) | HIV-infected Children on DTG-based ART (D3) | HIV-infected Children on LPV/R-based ART (L3) | HIV-uninfected Children (C3a) | HIV-uninfected Children (C3b)
Number analyzed (Participants) | 30 | 30 | 30 | 30 | 30
ng/mL | 243 [202 to 292] | 285 [224 to 363] | 491 [397 to 608] | 218 [175 to 272] | 272 [221 to 334]

5. Other Pre Specified Outcome: Cmax for Piperaquine in Single-dose Study
Description: Cmax for piperaquine: Maximal concentration in single-dose study to evaluate Safety
Time Frame: <24hr
Population: C1 and L1 were only for phase 1 safety evaluation, and those participants (n= 20 each arm) were not in phase 2 study,
Measure: Geometric Mean (95% Confidence Interval); unit: ng/mL
Groups:
- HIV-infected Children on LPV/R-based ART (L1): 20 HIV-infected children age 3 - 10 years on LPV/r-based ART for at least 10 days will take standard 3 consecutive once-daily oral doses of DP (20/120mg tablets) based on weight per 2015 WHO guidelines for DP. The brand name Duocotexin will be used.
  Dihydroartemisinin-piperaquine: It is expected that lopinavir/ritonavir (LPV/r) will increase DP exposure.
- HIV-uninfected Children (C1): 20 HIV-uninfected children age 3-10 years not on ART will take standard 3 consecutive once-daily oral doses of DP (20/120mg tablets) based on weight per 2015 WHO guidelines for DP. The brand name Duocotexin will be used. PK samples are collected after the 1st dose.
Arm/Group | HIV-infected Children on LPV/R-based ART (L1) | HIV-uninfected Children (C1)
Number analyzed (Participants) | 20 | 20
ng/mL | 96.3 [61.6 to 151] | 208 [145 to 299]

6. Other Pre Specified Outcome: AUC0-24h for Piperaquine in Single-dose Study
Description: AUC 0-24h (from time 0 to 24h) for piperaquine in single-dose study to evaluate safety.
Time Frame: 1 day
Population: Phase 1 study for safety evaluation was done with two arms (C1 and L1), and those participants (n= 20 each arm) were not in phase 2 study,
Measure: Geometric Mean (90% Confidence Interval); unit: hr.ug/mL
Arm/Group | HIV-infected Children on LPV/R-based ART (L1) | HIV-uninfected Children (C1)
Number analyzed (Participants) | 20 | 20
hr.ug/mL | 1.00 [0.73 to 1.37] | 1.89 [1.33 to 2.69]

7. Other Pre Specified Outcome: QTcF in Single-dose Safety Study
Description: Cardiotoxicity associated with PQ is QT interval prolongation. Electrocardiogram (ECG) will be performed to provide data on QT intervals in msec.
  Reported if QTcF>30ms
Time Frame: 28 days
Population: Single-dose study for safety evaluation was done with two arms (C1 and L1), and those participants (n= 20 each arm) were not in 3-dose full study,
Measure: Count of Participants; unit: Participants
Arm/Group | HIV-infected Children on LPV/R-based ART (L1) | HIV-uninfected Children (C1)
Number analyzed (Participants) | 20 | 20
Participants | 0 | 0

8. Other Pre Specified Outcome: The Association of Malnutrition and PK Exposure of DP in HIV-infected and HIV-uninfected Children
Description: Z-score is the anthropomorphic indicator of malnutrition measured as weight-for age (WFA). Children will be characterized as a) "stunted" but not underweight [i.e. weight for age (WFA) z-score>-2); b) underweight, but not stunted (WFA z-score ≤-2); or c) of normal nutritional status (WFA z-scores >-1).
Time Frame: 42 days
Reporting Status: Not Posted

9. Other Pre Specified Outcome: Assess Auto-induction of DHA From Single Dose to 3-doses
Description: DHA AUC0-8hr post the 1st dose is compared to AUC0-8hr post the 3rd dose
Time Frame: 3 days
Reporting Status: Not Posted

10. Other Pre Specified Outcome: CYP2B6 Pharmacogenetics and Its Impact on EFV PK
Description: To assess prevalence of CYP2B6 pharmacogenetic variants and their impact on EFV PK
Time Frame: 4 days
Reporting Status: Not Posted

11. Other Pre Specified Outcome: The Association of Anthropomorphic Indicators of Malnutrition Measured as Height-for-age (HFA) Z-score and PK Exposure of DP in HIV-infected and HIV-uninfected Children
Description: Children will be characterized as a) "stunted" but not underweight [i.e. height for age (HFA) z-score ≤-2); b) underweight, but not stunted (HFA z-score>-2); or c) of normal nutritional status (HFA z-scores >-1).
Time Frame: 42 days
Reporting Status: Not Posted

12. Other Pre Specified Outcome: The Effects of DP on EFV Pharmacokinetics as Measured by Trough-level (Cmin) of EFV
Description: Compare the trough EFV concentration on day 0 (pre-DP and EFV doses) to day 3 (24hr after DP and EFV doses)
Time Frame: 4 days
Reporting Status: Not Posted

13. Other Pre Specified Outcome: The Effects of DP on DTG Pharmacokinetics as Measured by Trough-level (Cmin) of DTG
Description: Pre-ART sample to quantify trough of DTG, sampled collected via venipuncture on Day 0, 2, & 3 to allow for comparisons of DTG level.
Time Frame: 4 days
Reporting Status: Not Posted

14. Other Pre Specified Outcome: The Effects of DP on LPV/r Pharmacokinetics as Measured by Trough-level (Cmin) of LPV/r
Description: Pre-ART sample to quantify trough of LPV/r, sampled collected via venipuncture on Day 0, 2, & 3 to allow for comparisons of LPV/r level.
Time Frame: 4 days
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 42 days
Groups:
- HIV-infected Children on LPV/R-based ART (L1): 20 HIV-infected children age 3 - 10 years on LPV/r-based ART for at least 10 days will take one oral dose DP (20/120mg tablets) based on weight per 2015 WHO guidelines for DP. The brand name Duocotexin will be used
  .
Arm/Group | HIV-infected Children on EFV-based ART (E3) | HIV-infected Children on DTG-based ART (D3) | HIV-infected Children on LPV/R-based ART (L3) | HIV-uninfected Children (C3a) | HIV-uninfected Children (C3b) | HIV-uninfected Children (C1) | HIV-infected Children on LPV/R-based ART (L1)
All-Cause Mortality (participants affected / at risk) | 0/30 | 0/30 | 0/30 | 0/30 | 0/30 | 0/20 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/30 | 0/30 | 0/30 | 0/30 | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 1/30 | 0/30 | 8/30 | 2/30 | 0/30 | 0/20 | 0/20
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | HIV-infected Children on EFV-based ART (E3) (N=30) | HIV-infected Children on DTG-based ART (D3) (N=30) | HIV-infected Children on LPV/R-based ART (L3) (N=30) | HIV-uninfected Children (C3a) (N=30) | HIV-uninfected Children (C3b) (N=30) | HIV-uninfected Children (C1) (N=20) | HIV-infected Children on LPV/R-based ART (L1) (N=20)
QTcF prolongation (Cardiac disorders) | 0 (0) | 0 (0) | 8 (8) | 2 (2) | 0 (0) | 0 (0) | 0 (0) — mild adverse QTcF changes of >30ms but less than 60ms
iron deficient anemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — moderate iron deficient anemia (low hemoglobin).

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-04-22): https://cdn.clinicaltrials.gov/large-docs/45/NCT04487145/Prot_SAP_000.pdf
  • Informed Consent Form (2022-04-07): https://cdn.clinicaltrials.gov/large-docs/45/NCT04487145/ICF_001.pdf